CLINICAL TRIAL: NCT02638454
Title: Role of MicroRNAs on Age and Contraction-induced Skeletal Muscle Growth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Roger A Fielding, Scientist II, Tufts University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 2860
Record Dates: First submitted 2015-12-17; First posted 2015-12-23 (Estimated); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Sarcopenia
Keywords: Exercise; Anabolic Resistance; Skeletal Muscle; microRNA
MeSH Terms: conditions — Sarcopenia; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- HL-YNG (Active Comparator): Healthy young sedentary males and females 20-30 yrs old
  Participants will undergo an acute bout of resistance exercise at 80% of their 1 repetition maximum (1RM, maximum strength) and will undergo muscle biopsies before, immediately after and 4 hours after the exercise.
  Interventions: Procedure: Acute Resistance Exercise
- FL-OLD (Experimental): Functionally-limited older sedentary males and females without sarcopenia (70-85 yrs old)
  Participants will undergo an acute bout of resistance exercise at 80% of their 1 repetition maximum (1RM, maximum strength) and will undergo muscle biopsies before, immediately after and 4 hours after the exercise.
  Interventions: Procedure: Acute Resistance Exercise
- SR-OLD (Experimental): Functionally-limited older sedentary males and females with clinically defined sarcopenia (70-85 yrs old)
  Participants will undergo an acute bout of resistance exercise at 80% of their 1 repetition maximum (1RM, maximum strength) and will undergo muscle biopsies before, immediately after and 4 hours after the exercise.
  Interventions: Procedure: Acute Resistance Exercise

INTERVENTIONS:
Procedure: Acute Resistance Exercise — 1 bout of high-intensity resistance exercise at 80% of the individuals 1 repetition maximum
  Other Names: Acute Strength Training

SUMMARY:
Sarcopenia is a predictor of functional-limitation, leading to loss of independence, lowered quality of life, and ultimately death. The impaired ability of aged skeletal muscle to adapt to anabolic stimulation may be a factor that contributes to sarcopenia. This project will provide novel insights into the role of microRNA in the attenuation of aging skeletal muscle to changes in gene expression after anabolic stimulation.

DETAILED DESCRIPTION:
The age-associated loss of skeletal muscle mass and function (sarcopenia) is associated with substantial social and economic costs. The plasticity and adaptability of skeletal muscle to contraction (ie. resistance-exercise) is a fundamental physiological event leading to larger and more robust skeletal muscle. However, muscle growth in response to resistance exercise (RE), like other anabolic stimuli, is attenuated in older adults. The cause of aberrant muscle adaptation with aging is complex. Recent work has revealed a novel role for small non-coding RNAs, called microRNAs (miRNA) in the regulation of gene expression. Using an integrated bioinformatics analysis of protein-coding gene and miRNA array data from young and older men, I identified ten specific miRNAs as important regulators of muscle plasticity (Plasticity Related miRs [PR-miRs]) leading to the transcriptional response to exercise and lean mass in young and older men. However, the precise mechanisms underlying the expression of PR-miRs on age-related changes in muscle anabolism and sarcopenia are currently unknown.

Thus, the overall objective of this K01 application will be to determine the mechanistic role(s) of these PR-miRs in skeletal muscle adaptation to anabolic stimulation in:

1. healthy young,
2. sarcopenic older and
3. age- and functionally-matched non-sarcopenic older males and females.

This will be accomplished by determine the differences in expression of PR-miRs with aging and sarcopenia in response to anabolic stimulation (AIM 1). Mechanistically determine the extent to which manipulation of PR-miR levels in vitro, in human primary myocytes, can reverse anabolic resistance observed with age and sarcopenia (AIM 2) and the effect of altering PR-miRs levels on skeletal muscle growth and development (AIM 3). This project will improve our understanding of the molecular mechanisms that contribute to the loss of skeletal muscle and eventually leading to the development of drug therapies for the treatment of sarcopenia in the ever growing aging population.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female
* 20-30 or 70-85 years of age
* Sedentary: Must not participate in any regular exercise sessions (participants who walk regularly or walk for exercise are eligible)
* Individuals must confirm good health
* BMI must be between 19-35 kg/m2
* Individuals must be fluent in English
* Willing to come to the HNRCA laboratory for study visits
* Short Physical Performance Battery of less than 9 (70-85 years of age cohort)
* 10 subjects with Normal Muscle Mass and 10 subjects with Low Muscle Mass as determined by DXA scan (70-85 years of age cohort) Low Muscle Mass is defined as Class I Sarcopenia, Skeletal Muscle Index within 1 to 2 standard deviations from the sex-specific mean of young adults

Exclusion Criteria:

* Lost or gained 7.5% or more of their body weight in the past 6 months
* Acute or terminal disease
* Significant immune disorder
* Types I and II Diabetes mellitus
* Uncontrolled hypertension (>180/100 mmHg)
* Neuromuscular disease
* Subjects must also not be participating in any regular endurance or resistance training exercise during the previous six months.
* Mini-mental state examination (MMSE) score of <23
* Because of the DXA scan and the unknown risk associated with the muscle biopsy procedure, women who are pregnant, planning to become pregnant, or are breastfeeding will be excluded from the study.

Subjects with a history of any of the following within the past 6 months will be excluded:

* Myocardial infarction in the past 6 months, or other symptomatic coronary artery disease.
* Surgery in previous 6 months
* Upper or lower extremity fracture in the previous 6 months
* Allergy to lidocaine

Subjects currently taking any of the following drugs or classes of drugs will be excluded:

* Anticoagulant therapy (Warfarin, Coumadin, or Plavix)
* ACE inhibitors
* Drugs that affects neuromuscular function
* Angiotensin receptor blockers
* Androgen or estrogen therapy or other hormone replacement therapy
* Low dose aspirin with known cardiovascular disease (e.g.: reported coronary artery disease, peripheral vascular disease, or previous stroke, or history of transient ischemic attacks)
* Diabetes medications (ie. metformin, insulin therapy, thiazolidinediones, sulfonylureas etc.)
* Chronic corticosteroid therapy

Laboratory blood test exclusions:

* Estimated GFR <30 mL/min/1.73m2
* Other abnormal screening lab values will be at the discretion of the study physician

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Change of microRNA expression in humans skeletal muscle after an acute bout of high intensity resistance exercise | Baseline, immediately (within 15-30 min after acute resistance exercise) and 4 hours after acute resistance exercise
  Determine if the expression of miRNA in skeletal muscle after an acute bout of high-intensity resistance exercise in young, functionally-limited older adults with and without low muscle mass

CONTACTS AND LOCATIONS:
Overall Officials: Donato A Rivas, PhD, Principal Investigator — Tufts University
Locations (1):
- Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided